CLINICAL TRIAL: NCT01780194
Title: Lumbar Fusion Compared With Conservative Treatment in Patients With Chronic Low Back Pain: a Meta-analysis
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: FUSION_META_TYH_2013
Record Dates: First submitted 2013-01-29; First posted 2013-01-30 (Estimated); Last update posted 2013-11-28 (Estimated); Status verified 2013-11

CONDITIONS: Comparison Between Effectiveness of Lumbar Fusion and Conservative Treatment

GROUPS / COHORTS (2):
- Lumbar fusion group
- Conservative treatment group

SUMMARY:
* To determine the effect size of lumbar fusion measured by Oswestry Disability Index and compared with conservative treatment in patients with chronic low back pain.
* Meta-analysis using fixed effect model synthesis method.
* Included studies were retrieved from Medline and Cochrane CENTRAL databases since 1990.

ELIGIBILITY:
Inclusion Criteria:

* controlled randomized or non-randomized studies

Exclusion Criteria:

* not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with chronic low back pain due to degenerative spinal conditions
Sampling Method: Probability Sample
Enrollment: 666 (Actual)
Dates: Start 2012-12; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Oswestry Disability Index | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Saltychev, PhD, Principal Investigator — Turku University Hospital

REFERENCES:
- [Derived] Saltychev M, Eskola M, Laimi K. Lumbar fusion compared with conservative treatment in patients with chronic low back pain: a meta-analysis. Int J Rehabil Res. 2014 Mar;37(1):2-8. doi: 10.1097/MRR.0b013e328363ba4b. PMID 23820296